CLINICAL TRIAL: NCT03066843
Title: A Randomized Controlled Trial Evaluating 5-aminolevulinic Acid Photodynamic Therapy With Different Incubation Times for the Treatment of Actinic Keratosis
Brief Title: Photodynamic Therapy Incubation Times for Actinic Keratosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00204459
Record Dates: First submitted 2017-02-24; First posted 2017-02-28 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid; Phototherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zero incubation with ALA (5-aminolevulinic acid) (Experimental): Subjects will receive zero time of incubation with ALA (5-aminolevulinic acid) before photodynamic blue light therapy.
  Interventions: Drug: ALA (5-aminolevulinic acid); Device: Blue light therapy
- One hour incubation with ALA (5-aminolevulinic acid) (Experimental): Subjects will receive one hour of incubation with ALA (5-aminolevulinic acid) before photodynamic blue light therapy.
  Interventions: Drug: ALA (5-aminolevulinic acid); Device: Blue light therapy

INTERVENTIONS:
Drug: ALA (5-aminolevulinic acid) — ALA (5-aminolevulinic acid) will be applied to subjects' skin for either zero time incubation or one hour incubation
  Other Names: Levulon kerastick
Device: Blue light therapy — Subjects will be exposed to blue light
  Other Names: BLU-U® Blue Light Photodynamic Therapy Illuminator

SUMMARY:
This is a randomized clinical trial evaluating blue light 5-aminolevulinic acid (ALA) photodynamic therapy with different incubation times for the treatment of actinic keratosis.

Subjects who are interested in participating, currently living in the Chicago metropolitan area, and meet inclusion and exclusion criteria will be enrolled in the study. Subjects will be randomized to either 1) zero time ALA incubation or 2) 1 hour ALA incubation. Demographic and health data will be collected prior to treatment initiation. Three visits will be conducted: screening, treatment, and follow up visit at 8 weeks.

This study is a pilot study designed to determine feasibility of this procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have been diagnosed with actinic keratosis.
2. Subjects who by the investigator deem to be suitable for photodynamic therapy of the face or scalp.
3. Males or females ≥ 18 years old
4. Fitzpatrick skin types I-VI
5. Subjects are in good health as judged by the investigator.
6. Subjects who are willing and have the ability to understand and provide informed consent for participation in the study and are able to communicate with the investigator.

Exclusion criteria:

1. Subjects who by the investigator are not suitable for photodynamic therapy.
2. Lesions suspicious or proven for skin cancer
3. History of 2 or more ALA- PDT treatments within the past 6 months.
4. Use of keratolytics within 2 days of initiation of treatment (e.g., >5% urea, glycolic acid, lactic acid, salicyclic acid)
5. Cryotherapy within the past 2 weeks.
6. Topical retinoids within the past 4 weeks
7. Procedures, such as microdermabrasion, ablative lasers, ALA-PDT, chemical peels, 5-fluorouraci, diclofenac, imiquimod within the past 8 weeks
8. Systemic retinoids within the past 6 months
9. Pregnant or breast feeding
10. Uncooperative subjects or subjects with neurological disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations.
11. Subjects who are unable to understand the protocol or give informed consent.
12. Subjects who in the opinion of the investigator are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in number of Actinic Keratosis (AK) lesions | Baseline and 8 Weeks
  The number of AK lesions will be counted by a live, blinded assessor at baseline and at Week 8 follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No